CLINICAL TRIAL: NCT04105192
Title: Randomized Controlled Clinical Trial on the Efficacy of a Natural Ingredient in Obesity in Subjects With a BMI Greater Than 25 kg / cm2
Brief Title: Effectiveness of a Natural Ingredient on Obesity
Acronym: (RACO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-0010
Record Dates: First submitted 2019-09-05; First posted 2019-09-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Overweight and Obesity; High Blood Pressure
MeSH Terms: conditions — Overweight; Obesity; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Lippia citriodora + sabdariffa) (Experimental): Consumption for 84 days of Lippia citriodora 325 mg + Hibiscus sabdariffa 175 mg.
  Two capsules per day will be consumed thirty minutes before breakfast orally for 84 days.
  Interventions: Dietary Supplement: dietary supplement consumption
- control group Placebo (sucrose) (Placebo Comparator): Consumption for 84 days of Lippia citriodora 325 mg + Hibiscus sabdariffa 175 mg or Placebo (sucrose) Two capsules per day will be consumed thirty minutes before breakfast orally for 84 days.
  Interventions: Dietary Supplement: dietary supplement consumption

INTERVENTIONS:
Dietary Supplement: dietary supplement consumption — Consumption of the product under study for 84 days, plecebo or experimental product

SUMMARY:
randomized, placebo-controlled clinical trial, with two parallel branches whose objective is to evaluate the efficacy of the product investigated on blood pressure and fat mass of subjects without pharmacotherapy.

DETAILED DESCRIPTION:
The subjects that meet the selection criteria will make a total of five visits to the research laboratory and will carry out the pre-established tests in the protocol. Subsequently, a statistical analysis will be carried out with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes with age between 18-65 years.
* Subjects with a body mass index greater than 25 and less than 35.
* Volunteers capable of understanding the clinical study and willing to comply with the procedures and requirements of the study.

Exclusion Criteria:

* Subjects under treatment that may affect body weight.
* Subjects with acute diseases.
* Volunteers with a history or presence of chronic pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunological, dermatological, urological, neurological, psychiatric, cardiovascular or pathology or malignant tumor disease.
* Subjects undergoing major surgery in the last 3 months.
* Subjects who quit smoking in the last 6 months or who intend to quit during the study.
* Subjects with allergies or eating disorders.
* Volunteers who are participating in another study that includes blood draws or dietary intervention.
* Pregnant or breastfeeding woman.
* Subjects whose condition does not make them eligible for the study, according to the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Total fat mass | From baseline to 84 days
  Dual X-ray absorptiometry (DEXA), measured in grams.
Fat mass in torso | From baseline to 84 days
  Dual X-ray absorptiometry (DEXA), measured in grams.
Fat mass in lower limbs | From baseline to 84 days
  Dual X-ray absorptiometry (DEXA), measured in grams.

SECONDARY OUTCOMES:
Fat mass | Time Frame: A record of body composition will be made five times during the 84 days of consumption. Measures will be taken at baseline, at 14 days, 28, 56 and 84 days. For this we will use a TANITA.
  Bioimpedancetry, in grams.
Muscle mass | Time Frame: A record of body composition will be made five times during the 84 days of consumption. Measures will be taken at baseline, at 14 days, 28, 56 and 84 days. For this we will use a TANITA.
  Bioimpedancetry, in grams.
Percentage of fat mass | Time Frame: A record of body composition will be made five times during the 84 days of consumption. Measures will be taken at baseline, at 14 days, 28, 56 and 84 days. For this we will use a TANITA.
  Bioimpedancetry.
blood samples: Glucidal metabolism and lipid metabolism. | Time Frame: Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of use.
  BASIC GLUCEMIA, TOTAL CHOLESTEROL, HDL CHOLESTEROL, LDL , CHOLESTEROL, TRIGLICERIDS, GLICATED HEMOGLOBIN. It was measured in milligrams per deciliter
Subjective sensation of product consumption | Time Frame: Subjects will complete the hedonic scale four times. at 14, 28, 56 and 84 days of consumption of the product under study.
  5-point hedonic scale. There are five points, being 1 I do not like and 5 I like it a lot. A scale will be passed through paper.
physical activity | Time Frame: An accelerometer will be placed twice on the subjects. The first time at baseline and the second after taking 84 days of consumption of the product under study
  MEASURED WITH ACTIGRAPH wGT3X-BT
liver safety variables | Hematological samples were taken before (day 0) and after consumption of the product (day 84) both in the control group and in the experimental group.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)
Weight | Time Frame: A record of body composition will be made five times during the 84 days of consumption. Measures will be taken at baseline, at 14 days, 28, 56 and 84 days. For these determinations we will use a scale (SECA).
  measured in Kg.
Height | Time Frame: A record of body composition will be made five times during the 84 days of consumption. Measures will be taken at baseline, at 14 days, 28, 56 and 84 days. For these determinations we will use a scale (SECA).
  Measured in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain